CLINICAL TRIAL: NCT06672016
Title: A Phase 3, Multicenter, Open-Label, Single-Arm Study of MR-130A-01 in Women of Childbearing Potential to Evaluate Contraceptive Efficacy and Safety
Brief Title: Study to Evaluate Contraceptive Efficacy and Safety of a Progestin Only Patch in Women of Childbearing Potential
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MR-130A-01-TD-3001
Record Dates: First submitted 2024-10-28; First posted 2024-11-04 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Female Contraception
Keywords: Female, Contraception, Progestin, Transdermal, Patch; Prevent Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- This is a single-arm study. (Experimental): The study patch is a transdermal system that contains the active ingredient progestin.
  This study is an open-label, single-arm study. This means that all participants in the study will receive the study patch
  Interventions: Drug: Transdermal system containing progestin

INTERVENTIONS:
Drug: Transdermal system containing progestin — MR-130A-01 transdermal system, patch to be used for female contraception

SUMMARY:
The Sponsor is developing a progestin-only contraceptive transdermal system (patch).

The main purpose of this study is to look at how safe the study patch is and how well it works in preventing pregnancy. The study will also look at how well the study patch is tolerated.

The study patch is a transdermal system that contains the active ingredient, progestin.

DETAILED DESCRIPTION:
Unintended pregnancy continues to be a significant reproductive health problem worldwide. Although the increase in the availability of longer-acting contraceptive methods has improved the situation, the continuing development of newer safe and effective contraception is crucial for women's health.

The development of a progestin-only contraceptive with more convenient dosing may provide women with additional options. The investigational patch is intended to provide an option for women who may not be able to use estrogen-containing combined hormonal contraceptives

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, post-menarcheal and premenopausal women at risk of pregnancy who are at least 16 years of age.
2. Desires to avoid pregnancy, is seeking to use hormonal contraception for at least 1 year.
3. Has negative UPT results at screening and at enrollment visits.
4. Has normal, regular menstrual cycles that are between 21 and 35 days in duration over the last 6 months.
5. Engages in regular heterosexual vaginal intercourse (at least once per cycle), with a partner who is not known to be sub fertile or infertile.
6. Agrees not to use other contraceptives or other methodology to prevent pregnancy during the study.
7. Able to understand and voluntarily provide written informed consent or assent (if the participant is adolescent prior to undergoing any trial related procedure) to participate in the study.

Exclusion Criteria:

1. Known or suspected pregnancy or planning pregnancy during next 12 months.
2. Participants with known hypersensitivity or intolerance to progestins, or any components of the progestin patch.
3. History or presence of dermal sensitivity to medicated patches or to topical applications including bandages, surgical tape.
4. Known infertility (current or known history) or history of sterilization in either partner.
5. Received injectable hormonal contraceptive therapy within 10 months of study enrollment.
6. Current use of hormonal contraceptive implants.
7. Has non-hormonal or hormonal intrauterine device (IUD) in place; or has had a recent IUD removal without one spontaneous menses after removal prior to the date of enrollment.
8. Recent surgical or medical abortion, miscarriage, ectopic pregnancy, or vaginal or cesarean delivery.
9. Participants lactating at the time of screening into the study or has occurrence of less than 3 regular menstrual cycles after cessation of lactation.
10. Anticipates routine use of condoms or any other form of back-up contraception for protection from sexually transmitted infections during the study or for emergency contraception.
11. Participants having a known contraindication to progestin-only contraception.
12. Known or suspected progestin sensitive malignant or premalignant conditions including but not limited to carcinoma of endometrium, ovary, or fallopian tubes.
13. Skin abnormality (e.g., tattoo or scar) at all possible application sites.
14. Long-term treatment with drugs or herbal products that are moderate/strong inducers or inhibitors of CYP3A4.
15. Has uncontrolled thyroid disorder (thyrotoxicosis or myxedema).
16. Has diagnosis of hereditary angioedema.
17. Participants with abnormal significant liver function tests as measured by liver function tests
18. Has a significantly abnormal cervical cancer screening test.
19. Participants with chlamydial or gonorrheal infection at screening.
20. Has unexplained vaginal bleeding within the past 6 months or any abnormal bleeding which is expected to recur during the study.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
To determine the contraceptive efficacy of progestin only patch when used over 13 cycles | 13 cycles [of 4 weeks (28 days)
  The primary efficacy endpoint will be pregnancy rate described by Pearl Index (PI). PI is defined as the number of pregnancies per 100 women-years.

SECONDARY OUTCOMES:
To determine the efficacy in obese population (Body mass index (BMI) ≥30.0 kg/m2) | 13 cycles [of 4 weeks (28 days)
  Assessment of PI in obese population (Body mass index (BMI) ≥30.0 kg/m2).
To determine the efficacy in non-obese population (Body mass index (BMI) <30.0 kg/m2) | 13 cycles [of 4 weeks (28 days)
  Assessment of PI in non-obese population (BMI <30.0 kg/m2).
Cycle-wise and cumulative pregnancy rates over 1 year | 13 cycles [of 4 weeks (28 days)
  Assessment of cycle-wise and cumulative pregnancy rates over 1 year using life table analysis.
Method failure PI | 13 cycles [of 4 weeks (28 days)
  Assessment of method failure PI.
Incidence of adverse events and serious adverse events | 13 cycles [of 4 weeks (28 days)
  Assessment of adverse events and serious adverse events.
Incidence of application site reactions | 13 cycles [of 4 weeks (28 days)
  Assessment of application site reactions.
Unscheduled bleeding | 13 cycles [of 4 weeks (28 days)
  Assessment of number of episode and days of unscheduled bleeding, proportion of participants reporting unscheduled bleeding.
Adhesion performance | 13 cycles [of 4 weeks (28 days)
  Assessment of patch adhesion performance as measured by 'Self-Reported Scoring System of Patch Adhesion Assessment Scale' Scores range from 0 to 4 where score 0 indicates the patch has essentially no lift off the skin and score 4 indicates the patch is detached and is completely off the skin.
progestin plasma concentrations | 5 cycles [of 4 weeks (28 days)
  Evaluation of progestin exposure in the subset of participants. PK samples for evaluation of progestin concentrations will be collected during cycles 2 and 5, for population PK and exposure-response analysis.

CONTACTS AND LOCATIONS:
Locations (51):
- United States (51):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - SEC Clinical Research, Dothan, Alabama
  - AMR Mobile, Mobile, Alabama
  - Velocity Clinical Research, Mobile, Alabama
  - Velocity Clinical Research, Phoenix, Arizona
  - Precision Trials, Phoenix, Arizona
  - Velocity Clinical Research Santa Ana, Huntington Park, California
  - Essential Access Health, Los Angeles, California
  - Women's Health Care Research Corp, San Diego, California
  - WR-Medical Center For Clinical Research, San Diego, California
  - AMR Fort Myers, Fort Myers, Florida
  - Altus Research, Lake Worth, Florida
  - OB GYN Associates of Mid Florida P.A., Leesburg, Florida
  - Genoma Research Group, Miami, Florida
  - Spotlight Research Center, Miami, Florida
  - New Age Med Research Corp, Miami, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Javarra and Privia Med, Savannah, Georgia
  - Leavitt ClinResearch, Idaho Falls, Idaho
  - Women's Healthcare Associates P.A., Idaho Falls, Idaho
  - AMR Newton, Newton, Kansas
  - AMR Lexington, Lexington, Kentucky
  - Clinical Trials Management, LLC, Covington, Louisiana
  - Velocity Clinical Research, Covington, Louisiana
  - Velocity Clinical Research, Lafayette, Louisiana
  - PraetorianPharmaResearch LLC, Marrero, Louisiana
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Velocity Clinical Research New Orleans, New Orleans, Louisiana
  - Valley OBGYN Clinic PC, Saginaw, Michigan
  - Alliance for Multispecialty Research, Kansas City, Missouri
  - Essential Women's Health, Las Vegas, Nevada
  - CenExel Hassman Research Institute, Marlton, New Jersey
  - Albuquerque Clinic Trials Inc, Albuquerque, New Mexico
  - Bosque Women's Care, Albuquerque, New Mexico
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Velocity Clinical Research, Beachwood, Ohio
  - Clinical Research Philadelphia, Philadelphia, Pennsylvania
  - Cedar Health Research, LLC, Euless, Texas
  - Helios Clinical Research, Fort Worth, Texas
  - ACRC Trials, Frisco, Texas
  - Javara, Houston, Texas
  - Clinical Trial Network LLC, Houston, Texas
  - Javara, Rowlett, Texas
  - Stephenville Medical and Surgical Clinic, Stephenville, Texas
  - Javara, Sugarland, Texas
  - Helios Clinical Research, Weatherford, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - AMR Norfolk, Norfolk, Virginia
  - Seattle Clinical Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No